CLINICAL TRIAL: NCT05659459
Title: The KIN-FAST Trial (KIN001 For Accelerated Symptoms Termination) A 4-week Double-blind, Randomized, Placebo-controlled, Phase II Study Evaluating the Effects of Oral Pamapimod 150 mg With Pioglitazone 10 mg Daily on COVID-19 Evolution and Recovery in Non-hospitalized Patients Infected With SARS-CoV-2 (Severe Acute Respiratory Syndrome-coronavirus-2)
Brief Title: The KIN-FAST Trial (KIN001 For Accelerated Symptoms Termination) in Non Hospitalized Patients Infected With SARS-CoV-2
Acronym: KIN-FAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor went bankrupt - trial was discontinued due to lack of financing
Sponsor: Kinarus AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIN001-204 - KIN-FAST
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KIN001 (Experimental): 75mg pamapimod oral tablet 5mg pioglitazone oral tablet twice daily for 14 days
  Interventions: Drug: KIN001
- Placebo (Placebo Comparator): 75mg pamapimod-placebo oral tablet 5mg pioglitazone-placebo oral tablet twice daily for 14 days
  Interventions: Drug: KIN001-Placebo

INTERVENTIONS:
Drug: KIN001 — Oral tablet
  Other Names: Combination Pamapimod 75mg with Pioglitazone 5mg
  Arms: KIN001
Drug: KIN001-Placebo — Comparator - Oral tablet with same appearance of KIN001
  Arms: Placebo

SUMMARY:
Clinical trial on safety and efficacy of KIN001 in non-hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized and placebo-controlled phase II trial to evaluate the safety and efficacy of KIN001 in non-hospitalized patients suffering from COVID-19. Randomization to one of two treatment arms (KIN001 versus Placebo) is at a ratio of 1:1.

Patients will receive treatment for 14 days and followed for another 14 days. The primary outcome is patient reported COVID-19 symptoms, using the FDA questionnaire developed for assessing COVID-19-related symptoms in outpatients.

The trial will be conducted in Switzerland and Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of symptomatic COVID-19 of less than 5 days' duration, with at least 1 point in at least 4 items of the symptom evaluation table, and at least 2 points in at least 2 items, OR a minimum total score of 6 points
2. Diagnosis of COVID-19 confirmed in the last 48 hours by a positive test for SARS-CoV-2 RNA by RT PCR or a rapid validated antigen test (excluding self-test), in a specimen from the upper respiratory tract, the saliva (antigen test), the lower respiratory tract or an expectorated sputum
3. No indication that the patient will be hospitalized in the next 48 hours for COVID-19 related reasons
4. Adult male or female patients aged ≥ 18 years
5. Females must have a negative pregnancy test or must be post-menopausal
6. Able to understand and willing to sign an IRB/IEC approved written informed consent document.
7. Able to understand and be available for daily phone calls to evaluate symptoms.

Exclusion Criteria:

1. Patients with an indication for hospitalization (e.g. SpO2 <92%)
2. Patients participating in another clinical trial with a new investigational drug or investigational non-drug treatment
3. Known allergy or intolerance to pamapimod or any other ingredient of the IMP or another P38 inhibitor
4. Known allergy or intolerance of clinical relevance to pioglitazone or any other ingredient of the IMP.
5. Patients where oral administration of pioglitazone is contraindicated (i.e. cardiac failure or history of cardiac failure (NYHA stages I to IV), with hepatic impairment, diabetic ketoacidosis, current bladder cancer or a history of bladder cancer, uninvestigated macroscopic haematuria
6. Any use of CYP450 2C8 inducers (e.g. rifampicin)
7. Known or suspected active viral (including HIV, hepatitis B, hepatitis C), bacterial, mycobacterial or fungal infection other than COVID-19. Virologic testing not required unless infection is suspected.
8. Pregnant or breastfeeding women
9. Any uncontrolled concurrent illness that would put the patient at a greater risk or limit compliance with the study requirements as determined at the discretion of the investigator
10. Liver enzyme elevation more than 3x above normal in the last 4 weeks or at inclusion
11. Patients who are detained or committed to an institution by a law court or by legal authorities (subject is vulnerable, such as deprived of freedom)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 symptoms evaluation | 28 days
  Number of days alive with no score > 1 in each of the symptoms and a maximum of 3 points in the total score*, measured from inclusion to day 28
  *Assessing COVID-19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment Guidance for Industry https://www.fda.gov/drugs/guidance-compliance-regulatory-information/guidances-drugs

SECONDARY OUTCOMES:
COVID-19 time to recovery | 28 days
  Time to clinical recovery, based on patient-reported daily evaluation of symptoms, and defined as the number of days from start of administration of the investigational agent to the first of two consecutive days when any symptoms scored as 2 or 3 at study entry are scored as 0-1 AND any symptoms scored as 0-1 at study entry are scored as 0
COVID-19 related hospital admissions | 28 days
  All-cause unplanned COVID-19 related hospital admissions
Safety and tolerability assessing treatment emergent adverse events | 28 days
  Safety and tolerability of KIN001
Total evaluation of COVID-10 symptoms score | 28 days
  Total sum of daily scores* of symptomes from inclusion to day 28
  *Assessing COVID-19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment Guidance for Industry https://www.fda.gov/drugs/guidance-compliance-regulatory-information/guidances-drugs

OTHER OUTCOMES:
Exploratory outcome - Sars-CoV-2 positive familiy members | 10 days
  Number of family members in the same household tested positive by Sars-CoV-2 PCR test two to 10 days after inclusion

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - Praxis am Ebertsplatz, Cologne
  - Velocity Clinical Research Hamburg, Hamburg
  - Praxis am Neckar, Heidelberg
- Switzerland (5):
  - Hôpital de la Tour, Meyrin
  - Cabinet Dr Clément, Nyon
  - Cabinet Dr. Thanh, Nyon
  - Cabinet Dr. Dang, Onex
  - Cabinet Dr. Schaller, Onex

IPD SHARING:
Plan to Share IPD: No
no IPD sharing plan